CLINICAL TRIAL: NCT04233853
Title: Improving Care for Patients with Depressive and Anxiety Disorders in Primary and Secondary Care: a Cluster-randomized Trial of a Consultation-liaison Intervention for General Practitioners
Brief Title: Consultation-Liaison Intervention for Patients with Depression and Anxiety in Primary Care
Acronym: CoLiPri
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Heidelberg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 407440_167436
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Depression; Anxiety
Keywords: Primary mental care; Collaborative care; Health services research; Common mental disorders; Implementation; Disease management
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CoLiPri intervention (Experimental): General practitioners and their screened patients have access to the consultation-liaison services for a total duration of 12 months, including standard screening, expert consultations, on demand patient referral for structured mental health diagnostics, psychoeducation and treatment planning, as well as brief psychotherapeutic intervention and triage.
  Interventions: Behavioral: CoLiPri intervention; Other: Usual primary care enhanced
- Usual primary care enhanced (Active Comparator): Usual primary care practice as offered in routine care. Enhanced means that practitioners receive a basic training which consists of guideline-based structured screening procedures for depression and anxiety mental disorders in primary care.
  Interventions: Other: Usual primary care enhanced

INTERVENTIONS:
Behavioral: CoLiPri intervention — General practitioners and their screened patients have access to the consultation-liaison services for a total duration of 12 months, including standard screening, expert consultations, on demand patient referral for structured mental health diagnostics, psychoeducation and treatment planning, as well as brief psychotherapeutic intervention and triage.
  Other Names: Consultation-liaison service
  Arms: CoLiPri intervention
Other: Usual primary care enhanced — Usual primary care practice as offered in routine care. Enhanced means that practitioners receive a basic training which consists of guideline-based structured screening procedures for depression and anxiety mental disorders in primary care.

SUMMARY:
The CoLiPri study is a cluster randomized controlled trial funded by the Swiss National Science Foundation to evaluate the clinical and cost effectiveness as well as the implementation of a complex consultation-liaison intervention to help improve symptoms of anxiety and depression of screened patients in primary care. The intervention includes expert consultations, on demand referral for structured mental health diagnostics, psychoeducation and treatment planning, as well as brief psychotherapeutic interventions and triage.

DETAILED DESCRIPTION:
Mental disorders such as depression or anxiety are serious and common health conditions that are highly prevalent in primary care. The primary care sector plays a key role in the treatment of common mental disorders as general practitioners (GPs) set the course for identification, diagnosis, therapy and referral to specialized treatment. The objectives of the CoLiPri study are to implement a complex consultation-liaison service at the intersection between primary and secondary care and to investigate its clinical and cost effectiveness in patients who are identified at primary care practices with elevated symptoms of depression and anxiety. Focus of the complex intervention is on improved collaboration and communication among GPs, mental health experts, and other services involved in the care of patients with common mental disorders. The novel service aims to support the decision-process at primary care practices, to increase access to evidence-based mental health treatment, and to help improve patients' pathways of care. The CoLiPri service for GPs include expert consultations, on-demand patient referral for structured diagnostics, and/or treatment planning, as well as brief psychotherapeutic interventions and triage. The effectiveness and cost effectiveness of the intervention as an add-on to enhanced usual primary care (usual care plus structured depression and anxiety screening) are evaluated in a cluster randomized clinical trial in screened patients with at least mild symptoms of depression and/or anxiety. In case of positive results, the service might serve as a model how to improve multi professional collaboration and clinical resource allocation for better delivery of mental health care.

ELIGIBILITY:
Inclusion Criteria:

* Patients scoring ≥5 on the PHQ-9 and/or scoring ≥5 on the GAD-7
* Presenting and treated at the participating practice
* Sufficient command of the German language
* Individual signed informed consent

Exclusion Criteria:

* Acute suicidality at the time of enrolment according to clinical evaluation
* A history of psychotic symptoms
* Bipolar Disorder Type-I or Type-II
* Acute substance-related and addictive disorder (i.e. as primary diagnosis)
* Severe cognitive impairment or other serious factors causing inability to follow the procedures of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2024-04-14 (Actual)

PRIMARY OUTCOMES:
Change in depressive and anxiety symptoms | Baseline, 3 months, 6 months
  Patient-reported depressive and anxiety symptoms will be assessed with the Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS) total score until 6-month follow-up. The PHQ-ADS combines the 9 items of the Depression Module of the PHQ (PHQ-9) and the 7 items of the General Anxiety Disorders 7 (GAD-7) to a single reliable and valid symptom measure. PHQ-ADS scores can range from 0 to 48 with higher scores indicating more severe depression/anxiety.

SECONDARY OUTCOMES:
Clinical response in depressive and anxiety symptoms | Baseline, 6 months
  Clinical response, defined as 50% reduction in patient-reported depressive and anxiety symptoms, will be assessed with the Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS) total score until 6-month follow-up.
Change in depressive and anxiety symptoms until 12-month follow-up | Baseline, 3 months, 6 months, 12 months
  Patient-reported depressive and anxiety symptoms will be assessed with the Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS) total score and subdomains, depression and anxiety, until 12-month follow-up.
Health-related quality of life | Baseline, 6 months, 12 months
  Health-related quality of life (HrQoL) and health state based on patient self-report assessed with the Short Form Health Survey SF-12 total and physical and mental health subscales until 6 and 12 months follow-up.
Health care utilization | Baseline, 6 months, 12 months
  Patients' self-reported health care utilization will be measured with the Client Sociodemographic and Service Receipt Inventory-German Version (CSSRI-D) as a basis for health economic analyses.
Utility-based health-related quality of life | Baseline, 3 months, 6 months, 12 months
  Utility-based health-related Quality of Life will be assessed via patient self-report with the five-level version of EQ-5D (EQ-5D-5L).
Cost-effectiveness | Baseline, 6 months, 12 months
  Cost-effectiveness evaluated with the information on healthcare utilization and productivity losses (direct and indirect costs) assessed with the CSSRI-D accumulated during 6 and 12 months. Quality-adjusted life years (QALYs) will be determined based on EQ-5D-5L based utility.

OTHER OUTCOMES:
Pathways of care | 12 months
  Healthcare utilization and pathways of care will be assessed based semi-standardized telephone interviews with the Longitudinal Interval Follow-Up Evaluation (LIFE) administered at 12-month follow-up.
Physician-patient relationship | Baseline, 6 months, 12 months
  The perceived quality of the physician-patient relationship will measured based on patient-self report with the German version of the Patient Reaction Assessment (PRA-D).
Patient satisfaction in primary care | 3 months, 6 months, 12 months
  The patients' satisfaction with GP treatment is assessed based on patient self-report with the Qualiskope-A.
Therapeutic alliance | Each session, approx. at 1 month, 2 months, 3 months, 4 months
  The therapeutic alliance is assessed after each individual CoLiPri session from the patient perspective with the German version of the Working Alliance Inventory-Short Revised (WAI-SR).
General self-esteem | Each session, approx. at 1 month, 2 months, 3 months, 4 months
  General self-esteem is measured with the revised version of the German Rosenberg Self-Esteem-Scale based patients self-report at each of the CoLiPri sessions within 12 months.
Quality of therapy sessions | Each session, approx. at 1 month, 2 months, 3 months, 4 months
  The quality of sessions delivered at the novel service will be monitored after each session within the 12 months with the patient version of the Bern Post Session Report (BPSR-P).
Client satisfaction | 3 months, 6 months, 12 months
  Client satisfaction with the CoLiPri services will be assessed in patients who have attended sessions based on patient self-report at 3-, 6-, and 12-month follow-up using the Fragebogen zur Messung der Patientenzufriedenheit (ZUF-8) which is the German version of the Client Satisfaction Questionnaire (CSQ-8).

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Watzke, Prof. Dr., Principal Investigator — University of Zurich; Markus Wolf, Dr., Principal Investigator — University of Zurich
Locations (1):
- University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Official website of the CoLiPri project (in German) — http://www.colipri.uzh.ch/de
- See also: Brief project description at the SNSF National Research Program 74 "Smarter Healthcare" — https://www.nfp74.ch/en/mpSTKsuFOIsU3w5B/project/project-watzke